CLINICAL TRIAL: NCT04848649
Title: Etude Pilote Exploratoire Des capacités Pronostiques de Rechute et Des Facteurs de Persistance de la mémoire Lymphocytaire T Dans Les Maladies Inflammatoires Chroniques
Brief Title: Shortening Treatments Of Chronic Inflammatory Conditions
Acronym: STOIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020/534
Record Dates: First submitted 2021-04-01; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Psoriasis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Psoriasis; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Other: Study arm

INTERVENTIONS:
Other: Study arm — Questionnaires, blood sample, skin (for psoriasis patients) or digestive (for IBD patients) biopsy and swab testing

SUMMARY:
Background Psoriasis is a common disease which is a source of major distress for patients and costs for the society. Treatments are effective but temporary and relapses occur, preferentially at sites previously involved. Locally, tissue resident memory T cells (TRM) cells prone to produce pathogenic cytokines accumulate in the outer layers of the resolved skin of psoriasis patients under treatment, and can trigger strong inflammatory responses upon reactivation, thus starting the cascade of the relapse. We have recently shown that the skin transcriptional responses after TRM cell activation in healed skin biopsies of patients could predict the time until the disease relapse. How to modify the local pool of TRM cells in the human skin is not known, but several factors leading to the establishment and the persistence of the TRM cells in the skin are suggested. First, the skin microbiota has emerged as a potent actor of the skin immunity, with the capacity to shape the pool of skin T cells in mice. Second, after TRM cells are settled in the skin, their lipid intake will impact their local survival. Last, in addition to these local factors, the gut subclinical inflammation that lead to bacterial translocation can trigger a more global state of inflammation in the body and could drive the local survival of the TRM cells in the skin.

Aims Our first aim in this project is to validate a tool to predict psoriasis relapse upon treatment withdrawal in a cohort of patients treated with systemic drugs- the STOPso cohort (Shortening Treatments Of Psoriasis). We will correlate the skin reaction to local TRM activation in resolved lesions to the time before relapse.

In parallel, we will characterize several factors likely to participate to the establishment, function and survival of the TRM cells in the skin. We will decipher the skin microbiota and mycobiota; the lipid composition of the outer layer of the skin; the presence of lipopolysaccharide in the blood, in order to better understand what factors should be targeted to modify the skin populations of TRM cells.

Methods Patients will be recruited through the Dermatology department of the university hospital of Besançon. We will use skin biopsies from resolved lesions to perform the characterization of the skin responses at the transcriptional level after local TRM activation with OKT-3 antibody compared to control. RNA will be analyzed with Nanostring technologies. For the microbiota analysis, we will use wet swabs and later DNA sequencing. The lipid composition and the circulating LPS will be analyzed after tape stripping, through the LabEx LipSTIC lipidomic platform of the region Bourgogne Franche-Comté. Patients will be followed up at Month 1, Month 6, Month 12 and Month 18 and at time of relapse if it occurs in between those intervals. Data about the disease activity (PASI, quality of life scores) and inter-current events will be registered at each time point.

Expected results and Perspectives The final aim of this project is to validate a tool available to clinicians to guide them in their decision to withdraw an efficient treatment in psoriasis, based on the skin reactivity to the resident T cells left locally after resolution of the inflammation. This would help reduce treatment length, and thus toxicities and costs to the health care systems. To open future perspectives, we also want to better understand the reasons why TRM populations tend to be retained in the skin, in order to develop remodeling strategies of the skin TRM populations.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis under systemic treatment for more than a year and in remission for at least 12 weeks: Physician Global Assessment [PGA] score 0-1, Psoriasis Area and Severity Index [PASI] score ≤ 3 OR inflammatory Bowel Disease [IBD] (Crohn's disease or ulcerative colitis) under systemic treatment for more than a year and in deep remission (clinical and endoscopic = SES CD 0-2 score for Crohn's, endoscopic Mayo score) in whom a de-escalation of treatment is scheduled.
* Agrrement of treatment discontinuation between patient and clinician before inclusion in this study.
* Informed Consent Form signed

Exclusion Criteria:

* Uncertain diagnosis
* Local immunomodulatory treatment for psoriasis ongoing or stopped for less than three weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Presence and activation of tissue-resident memory [TRM] lymphocytes | Month 6
  Assessment of predictive abilities of TRM lymphocytes in psoriasis relapse through transcriptomic analysis